CLINICAL TRIAL: NCT01187862
Title: Single-center, Randomized, Five-way Crossover Study to Investigate Low-dose Combinations of Caffeine, Efavirenz, Losartan, Omeprazole, Metoprolol, Chlorzoxazone and Midazolam ("Basel Cocktail") for Simultaneous Phenotyping of CYP1A2, CYP2B6, CYP2C9, CYP2C19, CYP2D6, CYP2E1 and CYP3A4 in Healthy Male Subjects
Brief Title: Pharmacokinetic Study to Investigate Low-dose Combinations of a Cocktail of Seven Drugs for Simultaneous Phenotyping of Cytochromes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: EKBB-94/10; 2010 DR 1136 (Other: Swissmedic)
Record Dates: First submitted 2010-08-23; First posted 2010-08-24 (Estimated); Last update posted 2015-04-17 (Estimated); Status verified 2015-04

CONDITIONS: Cytochrome; Pharmacokinetics
MeSH Terms: interventions — Caffeine; efavirenz; Losartan; Omeprazole; Metoprolol; Chlorzoxazone; Midazolam

ARMS (1):
- Basel cocktail (Other)
  Interventions: Drug: caffeine, efavirenz, losartan, omeprazole, metoprolol, chlorzoxazone and midazolam

INTERVENTIONS:
Drug: caffeine, efavirenz, losartan, omeprazole, metoprolol, chlorzoxazone and midazolam

SUMMARY:
The purpose of this study is to assess whether a cocktail of seven approved drugs (so-called "Basel cocktail") can be used for simultaneous phenotyping of CYP1A2, CYP2B6, CYP2C9, CYP2C19, CYP2D6, CYP2E1 and CYP3A4.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Male aged between 18 and 45 years
* No clinically significant findings on the physical examination
* Body mass index (BMI) between 18 and 28 kg/m2
* Systolic blood pressure (SBP) 100-145 mmHg, diastolic blood pressure (DBP) 50-90 mmHg, and heart rate (HR) 45-90 bpm (inclusive)
* 12-lead electrocardiogram (ECG) without clinically relevant abnormalities
* Hematology and clinical chemistry results not deviating from the normal range to a clinically relevant extent
* Negative results from urine drug screen
* Ability to communicate well with the investigator and to understand and comply with the requirements of the study

Exclusion Criteria:

* Known hypersensitivity to any excipients of the drug formulations
* Treatment with another investigational drug within 30 days prior to screening
* History or clinical evidence of alcoholism or drug abuse within the 3-year period prior to screening
* Excessive caffeine consumption, defined as mor than 800 mg per day
* History or clinical evidence of any disease and/or existence of any surgical or medical condition, which might interfere with the absorption, distribution, metabolism or excretion of the study drug
* Smoking within the last 3 months prior to screening
* Previous treatment with any prescribed or OTC medications (including herbal medicines such as St John's Wort) within 2 weeks prior to screening
* Loss of 250 ml or more of blood within 3 months prior to screening
* Any circumstances or conditions, which, in the opinion of the investigator, may affect full participation in the study or compliance with the protocol
* Legal incapacity or limited legal capacity at screening

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-07; Primary Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Assessment of phenotyping measures of seven drugs used as a cocktail

CONTACTS AND LOCATIONS:
Overall Officials: Manuel Haschke, MD, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital, Basel, Switzerland